CLINICAL TRIAL: NCT02357550
Title: Ketones Influence on Glucose Metabolism in Brain. A Human Positron Emission Tomography (PET) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: RM-1-10-72-106-14
Record Dates: First submitted 2015-01-26; First posted 2015-02-06 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2015-01

CONDITIONS: Ketone Body Metabolism; Brain Metabolism
MeSH Terms: interventions — Ketones

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Saline infusion. FDG-PET Scan. O2-PET scan. H2O-PET scan Muscle biopsy
  Interventions: Drug: placebo
- Hyperketonaemia (Experimental): Ketone infusion. FDG-PET Scan. O2-PET scan. H2O-PET scan Muscle biopsy
  Interventions: Drug: ketone

INTERVENTIONS:
Drug: ketone — 3-OHB is infused intravenously.
  Arms: Hyperketonaemia
Drug: placebo — Saline infusion.
  Arms: Control

SUMMARY:
This project tend to investigate the affection of ketone bodies on brain metabolism. This will be done by measuring human cerebral uptake of energy substrates, together with functional parameters, using PET imaging and appropriate radiotracers under hyperketonemia in healthy subjects by ketone infusion.

Hypotheses

1. Increased levels of ketone bodies in healthy subjects leads to decreased glucose uptake by brain cells contributing to hyperglycaemia.
2. Increased levels of ketone bodies in healthy subjects leads to increased cerebral blood flow.
3. Altered oxygen consumption during hyperketonemia in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* BMI 20-30 kg/m2

Exclusion Criteria:

* smoking
* alcohol abuse
* severe comorbidity
* blood donation 6 month prior
* claustrophobia

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Glucose metabolism in brain, CMR | t=240-360 minutes
  cerebral glucose metabolism measured by PET tracer during the above time frame

SECONDARY OUTCOMES:
Stress metabolism | 0-360 minutes
  growth hormone, cortisol, glucagon, adrenalin, ghrelin.
Oxygen use | T=150-200 minutes
  cerebral oxygen consumption measured by PET tracer during the above time frame
cerebral blood flow | t=180-250 minutes
  cerebral blood flow measured by PET tracer during the above time frame
Intramuscular signaling | t= 260 minutes
  protein and insulin signaling in muscle

CONTACTS AND LOCATIONS:
Overall Officials: Mads Svart, MD, Principal Investigator — Aarhus University / Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Lauritzen ES, Svart MV, Voss T, Moller N, Bjerre M. Impact of Acutely Increased Endogenous- and Exogenous Ketone Bodies on FGF21 Levels in Humans. Endocr Res. 2021 Feb;46(1):20-27. doi: 10.1080/07435800.2020.1831015. Epub 2020 Oct 19. PMID 33074729
- [Derived] Lauritsen KM, Sondergaard E, Svart M, Moller N, Gormsen LC. Ketone Body Infusion Increases Circulating Erythropoietin and Bone Marrow Glucose Uptake. Diabetes Care. 2018 Dec;41(12):e152-e154. doi: 10.2337/dc18-1421. Epub 2018 Oct 16. No abstract available. PMID 30327354